CLINICAL TRIAL: NCT00430248
Title: A Phase 3, Randomized, Multicenter, Double-Blind, Allopurinol-Controlled Study Assessing the Efficacy and Safety of Oral Febuxostat in Subjects With Gout.
Brief Title: Efficacy and Safety of Oral Febuxostat in Participants With Gout
Acronym: CONFIRMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F-GT06-153; U1111-1114-0226 (Registry Identifier: WHO)
Record Dates: First submitted 2007-01-25; First posted 2007-02-01 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Gout
Keywords: tophi; hyperuricemia; uric acid; Drug Therapy
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Febuxostat 40 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Febuxostat 80 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Allopurinol 200 mg or 300 mg QD (Active Comparator): (dependent on renal function)
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Febuxostat — Febuxostat 40 mg, capsules, orally, once daily for up to 6 months.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 40 mg QD
Drug: Febuxostat — Febuxostat 80 mg, capsules, orally, once daily for up to 6 months.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 80 mg QD
Drug: Allopurinol — Allopurinol 200 mg or 300 mg, capsules, orally, once daily for up to 6 months.
  Dose is dependent on the subject's renal function. Subjects with normal renal function or mild renal impairment received 300 mg once daily; subjects with moderate renal impairment received 200 mg once daily.
  Other Names: Zyloprim
  Arms: Allopurinol 200 mg or 300 mg QD

SUMMARY:
The purpose of this study is to compare the efficacy and safety of febuxostat, once Daily (QD), to allopurinol in subjects with hyperuricemia and gout.

DETAILED DESCRIPTION:
Renal impairment is common in subjects with gout, with the prevalence ranging from 50% to 70%. This population represents an unmet medical need as uricosuric drugs are contraindicated in these patients, and the only available treatment, allopurinol, may have to be dose reduced to avoid overt side effects.

Febuxostat (TMX-67) is a non-purine selective xanthine oxidase inhibitor being developed as an orally administered agent for management of hyperuricemia in patients with gout.

Treatment duration will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Has one or more of the American Rheumatism Association criteria for the diagnosis of gout.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Must have a serum urate level greater than or equal to 8.0 milligram per deciliter (mg/dL).

Exclusion Criteria:

* Have a severe, unstable, or life threatening medical condition that would likely prevent them from completing this study.
* Has a known body reaction to febuxostat, allopurinol, naproxen, any other non-steroidal anti-inflammatory drug (NSAID), aspirin, lansoprazole, colchicine, or any components in their formulation.
* History of xanthinuria.
* Alcohol consumption greater than 14/week.
* History of significant concomitant illness.
* Active liver or peptic ulcer disease.
* Has rheumatoid arthritis requiring treatment.
* Has estimated creatinine clearance less than 30 milliliter per minute (mL/min) calculated using the Cockcroft-Gault formula corrected for ideal body weight.
* Requires therapy with any other urate-lowering drug other than the study drug; long-term use of NSAIDs and COX-2 inhibitors; salicylates; thiazide diuretics; losartan; azathioprine; mercaptopurine; theophylline; intravenous (IV) colchicine; cyclosporine; cyclophosphamide; pyrazinamide; sulfamethoxazole;trimethoprim.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2269 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (258):
- United States (258):
  - Birmingham, Alabama
  - Hoover, Alabama
  - Hueytown, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Northport, Alabama
  - Ozark, Alabama
  - Tuscaloosa, Alabama
  - Chandler, Arizona
  - Gilbert, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sierra Vista, Arizona
  - Tucson, Arizona
  - Fort Smith, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Carmichael, California
  - Clovis, California
  - Concord, California
  - El Centro, California
  - Fair Oaks, California
  - Fullerton, California
  - Huntington Beach, California
  - Irvine, California
  - La Jolla, California
  - Laguna Hills, California
  - Los Angeles, California
  - Pasadena, California
  - Rancho Cucamonga, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - San Luis Obispo, California
  - Santa Barbara, California
  - Santa Maria, California
  - Torrance, California
  - Tustin, California
  - Vallejo, California
  - Vista, California
  - Walnut Creek, California
  - West Covina, California
  - Westlake Village, California
  - Whittier, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Highlands Ranch, Colorado
  - Littleton, Colorado
  - Longmont, Colorado
  - Wheat Ridge, Colorado
  - Danbury, Connecticut
  - Trumbull, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Boynton Beach, Florida
  - Brandon, Florida
  - Daytona Beach, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Gainsville, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Holly Hill, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Largo, Florida
  - Miami, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - New Smyrna Beach, Florida
  - Opa-locka, Florida
  - Orlando, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Haven, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Decatur, Georgia
  - Dunwoody, Georgia
  - Gainesville, Georgia
  - Marietta, Georgia
  - Stockbridge, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Meridian, Idaho
  - Nampa, Idaho
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Evanston, Illinois
  - Springfield, Illinois
  - Vernon Hills, Illinois
  - Elkhart, Indiana
  - Evansville, Indiana
  - Mishawaka, Indiana
  - Clive, Iowa
  - Des Moines, Iowa
  - Dubuque, Iowa
  - Kansas City, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Ruston, Louisiana
  - Shreveport, Louisiana
  - Slidell, Louisiana
  - Baltimore, Maryland
  - Frederick, Maryland
  - Owings Mills, Maryland
  - Prince Frederick, Maryland
  - Wheaton, Maryland
  - Fall River, Massachusetts
  - New Bedford, Massachusetts
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Stevensville, Michigan
  - Troy, Michigan
  - Chaska, Minnesota
  - Flowood, Mississippi
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Florissant, Missouri
  - Jefferson City, Missouri
  - Manchester, Missouri
  - Mexico, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Butte, Montana
  - Grand Island, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Dover, New Hampshire
  - Blackwood, New Jersey
  - Edison, New Jersey
  - Flemington, New Jersey
  - Manalapan, New Jersey
  - Medford, New Jersey
  - Midland Park, New Jersey
  - Albuquerque, New Mexico
  - Endwell, New York
  - Mineola, New York
  - New York, New York
  - Smithtown, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Harrisburg, North Carolina
  - High Point, North Carolina
  - Lenoir, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Austintown, Ohio
  - Beachwood, Ohio
  - Chardon, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Hudson, Ohio
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Perrysburg, Ohio
  - Toledo, Ohio
  - Willoughby Hills, Ohio
  - Youngstown, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Eugene, Oregon
  - Lake Oswego, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - East Norriton, Pennsylvania
  - Feasterville-Trevose, Pennsylvania
  - Harrisburg, Pennsylvania
  - Lansdale, Pennsylvania
  - Mechanicsburg, Pennsylvania
  - Morrisville, Pennsylvania
  - Penndel, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Scotland, Pennsylvania
  - West Reading, Pennsylvania
  - Cranston, Rhode Island
  - East Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Orangeburg, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Clarksville, Tennessee
  - Collierville, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - New Tazewell, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Bellaire, Texas
  - Bryan, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Killeen, Texas
  - Lake Jackson, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Waco, Texas
  - Layton, Utah
  - Midvale, Utah
  - Salt Lake City, Utah
  - St. George, Utah
  - West Jordan, Utah
  - Chesapeake, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Everett, Washington
  - Gig Harbor, Washington
  - Lakewood, Washington
  - Olympia, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - Monroe, Wisconsin
  - Oregon, Wisconsin

REFERENCES:
- [Result] Becker MA, Schumacher HR, Espinoza LR, Wells AF, MacDonald P, Lloyd E, Lademacher C. The urate-lowering efficacy and safety of febuxostat in the treatment of the hyperuricemia of gout: the CONFIRMS trial. Arthritis Res Ther. 2010;12(2):R63. doi: 10.1186/ar2978. Epub 2010 Apr 6. PMID 20370912
- [Result] Wortmann RL, Macdonald PA, Hunt B, Jackson RL. Effect of prophylaxis on gout flares after the initiation of urate-lowering therapy: analysis of data from three phase III trials. Clin Ther. 2010 Dec;32(14):2386-97. doi: 10.1016/j.clinthera.2011.01.008. PMID 21353107
- [Result] Becker MA, MacDonald PA, Hunt B, Gunawardhana L. Treating hyperuricemia of gout: safety and efficacy of febuxostat and allopurinol in older versus younger subjects. Nucleosides Nucleotides Nucleic Acids. 2011 Dec;30(12):1011-7. doi: 10.1080/15257770.2011.603715. PMID 22132950
- [Result] Chohan S, Becker MA, MacDonald PA, Chefo S, Jackson RL. Women with gout: efficacy and safety of urate-lowering with febuxostat and allopurinol. Arthritis Care Res (Hoboken). 2012 Feb;64(2):256-61. doi: 10.1002/acr.20680. PMID 22052584
- [Derived] Becker MA, MacDonald PA, Hunt BJ, Jackson RL. Diabetes and gout: efficacy and safety of febuxostat and allopurinol. Diabetes Obes Metab. 2013 Nov;15(11):1049-55. doi: 10.1111/dom.12135. Epub 2013 Jun 12. PMID 23683134
- [Derived] Jackson RL, Hunt B, MacDonald PA. The efficacy and safety of febuxostat for urate lowering in gout patients >/=65 years of age. BMC Geriatr. 2012 Mar 21;12:11. doi: 10.1186/1471-2318-12-11. PMID 22436129
- [Derived] Wells AF, MacDonald PA, Chefo S, Jackson RL. African American patients with gout: efficacy and safety of febuxostat vs allopurinol. BMC Musculoskelet Disord. 2012 Feb 9;13:15. doi: 10.1186/1471-2474-13-15. PMID 22316106
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 324 sites in the United States from 16 February 2007 to 12 March 2008.
Pre-assignment Details: Subjects who were currently receiving urate-lowering therapy discontinued those urate-lowering therapies and initiated prophylactic medications before enrollemnt in once daily (QD) treatment groups.
Groups:
- Febuxostat 40 mg QD: Febuxostat 40 mg, orally, once daily for up to 6 months.
- Febuxostat 80 mg QD: Febuxostat 80 mg, orally, once daily for up to 6 months.
- Allopurinol 200 mg or 300 mg QD: Allopurinol, orally, for up to 6 months. Dose of allopurinol received was based on renal status. Subjects with normal renal function or mild renal impairment received 300 mg QD; subjects with moderate renal impairment received 200 mg QD.
Period: Overall Study
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Started | 757 | 756 | 756
Completed | 632 | 598 | 621
Not Completed | 125 | 158 | 135
Not completed — Adverse Event | 49 | 61 | 64
Not completed — Protocol Violation | 10 | 2 | 4
Not completed — Personal Reasons | 12 | 24 | 9
Not completed — Lost to Follow-up | 28 | 33 | 28
Not completed — Therapeutic Failure | 1 | 1 | 1
Not completed — Withdrawal by Subject | 14 | 20 | 16
Not completed — Inclusion/Exclusion Criteria Not Met | 0 | 2 | 0
Not completed — Gout Flare | 3 | 7 | 2
Not completed — Reason Not Specified | 8 | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD | Total
Number analyzed (Participants) | 757 | 756 | 756 | 2269
Age, Customized [Number; unit: subjects]
  <45 years of age | 192 | 196 | 180 | 568
  45 to <65 years of age | 450 | 432 | 445 | 1327
  ≥65 years of age | 115 | 128 | 131 | 374
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.68) | 53.0 (11.79) | 52.9 (11.73) | 52.8 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 46 | 47 | 128
  Male | 722 | 710 | 709 | 2141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 49 | 53 | 149
  Not Hispanic or Latino | 710 | 707 | 702 | 2119
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 10 | 6 | 22
  Asian | 26 | 25 | 37 | 88
  Native Hawaiian or Other Pacific Islander | 11 | 10 | 11 | 32
  Black or African American | 83 | 78 | 67 | 228
  White | 620 | 618 | 625 | 1863
  More than one race | 11 | 15 | 8 | 34
  Unknown or Not Reported | 0 | 0 | 2 | 2
Body Mass Index [Number; unit: subjects]
  <18.5 kilograms per meter² (kg/m²) | 0 | 1 | 1 | 2
  18.5 kg/m² to <25 kg/m² | 50 | 46 | 42 | 138
  25 kg/m² to <30 kg/m² | 215 | 232 | 236 | 683
  ≥30 kg/m² | 490 | 476 | 476 | 1442
  Missing | 2 | 1 | 1 | 4
Cardiovascular Disease [Number; unit: subjects]
  No | 336 | 316 | 320 | 972
  Yes | 421 | 440 | 436 | 1297
Renal Function [Number; unit: subjects] — Moderate renal impairment - baseline estimated creatinine clearance (CLcr) 30 milliliters per minute (mL/min) to 59 mL/min; Mild renal impairment - baseline estimated CLcr 60 mL/min to 89 mL/min; Normal renal function - estimated CLcr ≥90 mL/min.
  CLcr calculated using the Cockroft-Gault formula corrected for ideal body weight.
  subjects
    Moderate Renal Impairment | 130 | 136 | 136 | 402
    Mild Renal Impairment | 349 | 367 | 365 | 1081
    Normal Renal Function | 278 | 253 | 255 | 786
Mean Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 32.9 (6.37) | 32.9 (6.39) | 32.7 (6.23) | 32.8 (6.33)
Serum Urate [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 9.6 (1.15) | 9.6 (1.20) | 9.5 (1.19) | 9.6 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Whose Serum Urate Level is <6.0 Milligrams Per Deciliter (mg/dL) at the Final Visit.
Description: The percentage of subjects whose serum urate level was <6.0 mg/dL at the Final Visit was summarized. The Final Visit was the last visit at which a serum urate value was collected.
Time Frame: Last Visit on treatment (up to 6 months)
Population: Analysis was performed on intent-to-treat (ITT) subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had baseline serum urate ≥8.0 mg/dL. A subject's baseline value was used in the primary analysis if no postbaseline serum urate level was obtained.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 757 | 756 | 755
percentage of subjects | 45.2 | 67.1 | 42.1
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; The primary comparison was between febuxostat 40 mg and allopurinol treatment groups; Test type: Non-Inferiority or Equivalence — Noninferiority of febuxostat 40 mg to allopurinol was declared if the value of the lower bound of the 95% confidence interval for the difference was greater than -10%; Difference in percentage = 3.1, 95% CI [-1.9 to 8.1]
Statistical Analysis 2: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.233, Fisher Exact — The test for superiority was performed using Fisher's exact test (two-tailed 0.05 significance level)
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Comparisons between treatment groups were performed using Fisher's exact test (two-tailed 0.05 significance level); Difference in percentage = 24.9, 95% CI [20.1 to 29.8]
Statistical Analysis 4: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Comparisons between treatment groups were performed using Fisher's exact test (two-tailed 0.05 significance level); Difference in percentage = 21.9, 95% CI [17.0 to 26.8]

2. Secondary Outcome: Percentage of Renal Impairment Subjects Whose Final Visit Serum Urate Level is <6.0 mg/dl
Description: The percentage of subjects with mild-to-moderate renal impairment whose serum urate was <6.0 mg/dL at the final visit was summarized. The final visit was the last visit at which a serum urate value was collected.
Time Frame: Last Visit on treatment (up to 6 months)
Population: Analysis was performed on the ITT subjects with mild-to-moderate renal impairment (estimated creatinine clearance of 30 mL/min to 89 mL/min), with a post-baseline serum urate level.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 479 | 503 | 501
percentage of subjects | 49.7 | 71.6 | 42.3
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.021, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

3. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <6.0 mg/dL at Month 2 Visit.
Description: Serum urate values were obtained at the Month 2 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 2 visit was summarized.
Time Frame: Month 2
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 2 visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 703 | 691 | 685
percentage of subjects | 49.1 | 74.1 | 43.2
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.031, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

4. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <6.0 mg/dL at Month 4 Visit.
Description: Serum urate values were obtained at the Month 4 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 4 visit was summarized.
Time Frame: Month 4
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 4 visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 652 | 636 | 646
percentage of subjects | 47.1 | 75.2 | 45.5
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.578, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

5. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <6.0 mg/dL at Month 6 Visit.
Description: Serum urate values were obtained at the Month 6 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 6 visit was summarized.
Time Frame: Month 6
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 6 visit.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 618 | 596 | 616
percentage of participants | 48.9 | 75.3 | 46.6
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.426, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

6. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <5.0 mg/dL at Month 2 Visit.
Description: Serum urate values were obtained at the Month 2 visit. The percentage of subjects whose serum urate was <5.0 mg/dL at the Month 2 visit was summarized.
Time Frame: Month 2
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 2 visit
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 703 | 691 | 685
percentage of subjects | 15.4 | 45.9 | 11.7
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.050, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

7. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <5.0 mg/dL at Month 4 Visit.
Description: Serum urate values were obtained at the Month 4 visit. The percentage of subjects whose serum urate was <5.0 mg/dL at the Month 4 visit was summarized.
Time Frame: Month 4
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 4 visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 652 | 636 | 646
percentage of subjects | 15.0 | 51.6 | 13.5
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.428, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

8. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <5.0 mg/dL at Month 6 Visit.
Description: Serum urate values were obtained at the Month 6 visit. The percentage of subjects whose serum urate was <5.0 mg/dL at the Month 6 visit was summarized.
Time Frame: Month 6
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 6 visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 618 | 596 | 616
percentage of subjects | 19.3 | 49.7 | 14.8
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.041, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

9. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <5.0 mg/dL at Final Visit.
Description: The percentage of subjects whose serum urate level was <5.0 mg/dL at the Final Visit was summarized. The Final Visit was the last visit at which a serum urate values was collected.
Time Frame: Last Visit on treatment (up to 6 months)
Population: Analysis was performed on the ITT subjects with a post-baseline serum urate value.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 757 | 756 | 755
percentage of subjects | 16.5 | 44.0 | 13.2
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.083, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

10. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <4.0 mg/dL at Month 2 Visit
Description: Serum urate values were obtained at the Month 2 visit. The percentage of subjects whose serum urate was <4.0 mg/dL at the Month 2 visit was summarized.
Time Frame: Month 2
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 2 visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 703 | 691 | 685
percentage of subjects | 2.1 | 17.5 | 1.5
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.421, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

11. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <4.0 mg/dL at Month 4 Visit
Description: Serum urate values were obtained at the Month 4 visit. The percentage of subjects whose serum urate was <4.0 mg/dL at the Month 4 visit was summarized.
Time Frame: Month 4
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 4 visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 652 | 636 | 646
percentage of subjects | 2.0 | 18.6 | 1.4
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.520, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

12. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <4.0 mg/dL at Month 6 Visit
Description: Serum urate values were obtained at the Month 6 visit. The percentage of subjects whose serum urate was <4.0 mg/dL at the Month 6 visit was summarized.
Time Frame: Month 6
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 6 visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 618 | 596 | 616
percentage of subjects | 3.1 | 20.3 | 1.8
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.195, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

13. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <4.0 mg/dL at Final Visit
Description: The percentage of subjects whose serum urate level was <4.0 mg/dL at the Final Visit was summarized. The Final Visit was the last visit at which a serum urate values was collected.
Time Frame: Last Visit on treatment (up to 6 months)
Population: Analysis was performed on the ITT subjects with a post-baseline serum urate value.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 757 | 756 | 755
percentage of subjects | 2.5 | 17.5 | 1.5
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.196, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — The a priori threshold for statistical significance was 0.05 (two-tailed)

14. Secondary Outcome: Mean Percent Change From Baseline in Serum Urate Levels at Month 2 Visit.
Description: Serum urate values were obtained at the Month 2 visit. The percent change in serum urate from baseline to the Month 2 visit was summarized.
Time Frame: Baseline and Month 2
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 2 visit.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 703 | 691 | 685
percent change from baseline | -35.1 (12.8) | -44.5 (15.5) | -33.8 (13.2)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.079, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level

15. Secondary Outcome: Mean Percent Change From Baseline in Serum Urate Levels at Month 4 Visit
Description: Serum urate values were obtained at the Month 4 visit. The percent change in serum urate from baseline to the Month 4 visit was summarized.
Time Frame: Baseline and Month 4
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 4 visit.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 652 | 636 | 646
percent change from baseline | -34.9 (13.1) | -45.5 (15.6) | -34.5 (12.8)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.685, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level

16. Secondary Outcome: Mean Percent Change From Baseline in Serum Urate Levels at Month 6 Visit.
Description: Serum urate values were obtained at the Month 6 visit. The percent change in serum urate from baseline to the Month 6 visit was summarized.
Time Frame: Baseline and Month 6
Population: Analysis was performed on the ITT subjects with a serum urate value at Month 6 visit.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 618 | 596 | 616
percent change from baseline | -35.6 (13.2) | -45.1 (16.0) | -34.4 (13.3)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.153, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level

17. Secondary Outcome: Mean Percent Change From Baseline in Serum Urate Levels at Final Visit.
Description: The percent change in serum urate from baseline to the Final visit was summarized. The final visit was the last visit at which a serum urate value was collected.
Time Frame: Baseline and Last Visit on treatment (up to 6 months)
Population: Analysis was performed on the ITT subjects with a post-baseline serum urate value.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Number analyzed (Participants) | 757 | 756 | 755
percent change from baseline | -33.1 (15.5) | -40.6 (19.9) | -31.3 (16.2)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p = 0.050, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Allopurinol 200 mg or 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level
Statistical Analysis 3: Comparison: Febuxostat 40 mg QD vs Febuxostat 80 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is from contrast within the framework of the ANOVA with significance at the 0.05 level

ADVERSE EVENTS:
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Serious Adverse Events (participants affected / at risk) | 19 | 28 | 31
Other Adverse Events (participants affected / at risk) | 193 | 167 | 166
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Leukocytoses not elsewhere classified (NEC) (Blood and lymphatic system disorders) | 0/757 | 1/756 | 0/756
Thrombocytopenias (Blood and lymphatic system disorders) | 0/757 | 1/756 | 0/756
Cardiac Conduction Disorders (Cardiac disorders) | 0/757 | 2/756 | 0/756
Cardiac Hypertensive Complications (Cardiac disorders) | 0/757 | 0/756 | 1/756
Coronary Artery Disorders NEC (Cardiac disorders) | 2/757 | 0/756 | 2/756
Heart Failures NEC (Cardiac disorders) | 2/757 | 0/756 | 1/756
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 1/757 | 2/756 | 1/756
Supraventricular Arrhythmias (Cardiac disorders) | 0/757 | 1/756 | 0/756
Inner Ear Signs and Symptoms (Ear and labyrinth disorders) | 0/757 | 1/756 | 0/756
Acute and Chronic Pancreatitis (Gastrointestinal disorders) | 0/757 | 1/756 | 0/756
Benign Neoplasms GastrointestinaI (Excluding Oral Cavity) (Gastrointestinal disorders) | 1/757 | 0/756 | 0/756
Dyspeptic Signs and Symptoms (Gastrointestinal disorders) | 0/757 | 0/756 | 1/756
Gastrointestinal & Abdominal Pains (Excluding Oral and Throat) (Gastrointestinal disorders) | 0/757 | 0/756 | 1/756
Gastrointestinal Ulcers and Perforation, Site Unspecified (Gastrointestinal disorders) | 0/757 | 0/756 | 1/756
Intestinal Haemorrhages (Gastrointestinal disorders) | 0/757 | 0/756 | 1/756
Intestinal Ulcers and Perforation NEC (Gastrointestinal disorders) | 2/757 | 1/756 | 0/756
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 0/757 | 0/756 | 1/756
Non-Site Specific Gastrointestinal Haemorrhages (Gastrointestinal disorders) | 0/757 | 1/756 | 0/756
General Signs and Symptoms NEC (General disorders) | 1/757 | 0/756 | 0/756
Pain and Discomfort NEC (General disorders) | 1/757 | 2/756 | 1/756
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 0/757 | 0/756 | 3/756
Allergies to Food, Food Additives, Drugs and Other Chemicals (Immune system disorders) | 0/757 | 0/756 | 1/756
Anaphylactic Responses (Immune system disorders) | 1/757 | 0/756 | 0/756
Abdominal and Gastrointestinal Infections (Infections and infestations) | 2/757 | 0/756 | 1/756
Bacterial Infections NEC (Infections and infestations) | 1/757 | 1/756 | 2/756
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 1/757 | 1/756 | 3/756
Sepsis, Bacteraemia, Viraemia, and Infections (Infections and infestations) | 0/757 | 1/756 | 1/756
Fractures and Dislocations NEC (Injury, poisoning and procedural complications) | 0/757 | 1/756 | 0/756
Muscle, Tendon and Ligament Injuries (Injury, poisoning and procedural complications) | 0/757 | 1/756 | 0/756
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 0/757 | 2/756 | 0/756
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 1/757 | 0/756 | 1/756
Upper limb Fractures and Dislocations (Injury, poisoning and procedural complications) | 0/757 | 1/756 | 1/756
Purine Metabolism Disorders NEC (Metabolism and nutrition disorders) | 0/757 | 1/756 | 1/756
Total Fluid Volume Decreased (Metabolism and nutrition disorders) | 1/757 | 0/756 | 0/756
Joint Related Disorders NEC (Musculoskeletal and connective tissue disorders) | 0/757 | 1/756 | 0/756
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 0/757 | 1/756 | 0/756
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 0/757 | 1/756 | 0/756
Bladder Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/757 | 1/756 | 0/756
Breast and Nipple Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/757 | 0/756 | 0/756
Colonic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/757 | 0/756 | 1/756
Nervous System Neoplasms Unpecified Malignancy NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/757 | 0/756 | 1/756
Nonsmall Cell Neoplasm Malignant/Respiratory Type Specified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/757 | 0/756 | 1/756
Prostatic Neoplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/757 | 1/756 | 0/756
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/757 | 1/756 | 3/756
Central Nervous System Hemorrhages & Cerebrovascular Accidents (Nervous system disorders) | 0/757 | 1/756 | 1/756
Disturbances in Consciousness NEC (Nervous system disorders) | 0/757 | 0/756 | 3/756
Increased Intracranial Pressure Disorders (Nervous system disorders) | 0/757 | 1/756 | 0/756
Neurological Signs and Symptoms NEC (Nervous system disorders) | 1/757 | 0/756 | 0/756
Transient Cerebrovascular Events (Nervous system disorders) | 1/757 | 1/756 | 1/756
Renal Failure and Impairment (Renal and urinary disorders) | 0/757 | 1/756 | 0/756
Renal Vascular and Ischaemic Conditions (Renal and urinary disorders) | 0/757 | 1/756 | 0/756
Prostatic Signs, Symptoms and Disorders NEC (Reproductive system and breast disorders) | 0/757 | 1/756 | 0/756
Bronchospasms and Obstruction (Respiratory, thoracic and mediastinal disorders) | 0/757 | 1/756 | 1/756
Pulmonary Thrombotic and Embolic Conditions (Respiratory, thoracic and mediastinal disorders) | 0/757 | 1/756 | 0/756
Aortic Aneurysms and Dissections (Vascular disorders) | 1/757 | 0/756 | 1/756
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 200 mg or 300 mg QD
Upper Respiratory Tract Infections (Infections and infestations) | 71/757 | 53/756 | 57/756
Liver Function Analyses (Investigations) | 63/757 | 52/756 | 50/756
Diarrhoea (Excluding Infective) (Gastrointestinal disorders) | 45/757 | 47/756 | 57/756
Musculoskeletal and Connective Tissues Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 43/757 | 38/756 | 32/756

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.